CLINICAL TRIAL: NCT01107314
Title: Vasopressin Deficiency in Hemorrhagic Shock
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0528-H; A-13969.2 (Other Grant/Funding Number: DoD)
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2012-03

CONDITIONS: Body Response to Trauma
MeSH Terms: interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- trauma patient: SBP less than 90mmHg
  Interventions: Other: Phlebotomy

INTERVENTIONS:
Other: Phlebotomy — Blood draws (total 48 cc blood)

SUMMARY:
In this study we hope to delineate the typical vasoactive mediator response of trauma patients to shock. We plan to assess serum levels of vasopressin and also catecholamines, angiotensin, and cortisol during resuscitation of trauma patients to delineate high risk populations for vasopressin deficiency.

DETAILED DESCRIPTION:
This is a prospective observational study. The only research-driven procedure will be the removal of blood samples at designated time points(total blood removed 48 cc per patient). Hemodynamic, fluid infusion and agitation/pain data (RAMSEY Score) will prospectively be collected for research purposes. We will collect data from a convenience sample of patients (when research staff is available) over a one year period.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male or female patient presumed to be at least 18 years of age;
* Patient has a reported or actual systolic blood pressure < 90 mmHg within 1 hour of arrival to the Emergency Room;
* Patient has clinical evidence of acute traumatic injury;

Exclusion Criteria:

* Patient is asystolic or requires CPR prior to arrival;
* Patient was transferred from an outside facility
* Patient known to be pregnant
* Patient known to be prisoner

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: observational study - trauma patients admitted to University Hospital
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04-30 (Actual); Study Completion 2011-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Cohn, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- UTHSCSA, San Antonio, Texas, United States